CLINICAL TRIAL: NCT03305094
Title: The Effect of Remote Ischemic Preconditioning in Aortic Valve Replacement Surgery : a Randomized Controlled Trial
Brief Title: The Effect of Remote Ischemic Preconditioning in Aortic Valve Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Pierre Voisine, Cardiac surgeon, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONDOR-21082
Record Dates: First submitted 2017-09-28; First posted 2017-10-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Stenosis; Cardiopulmonary Bypass
Keywords: Remote ischemic preconditioning; Myocardial infarction; Cardiac surgery
MeSH Terms: conditions — Aortic Valve Stenosis; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective trial
Who Masked: Participant
Masking Description: Participant is blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Sham remote ischemic preconditioning on the right arm is induced with a blood pressure cuff inflation at 20 mm Hg for 5 min and followed by a 5 min reperfusion at 0 mm Hg. The sham ischemia-reperfusion cycle is performed 3 times for a total of 30 min. This procedure is done after anesthetic induction, but before the patient is placed on cardiopulmonary bypass.
  A 20 mm Hg blood pressure cuff on the right arm does not induce ischemia.
  Interventions: Procedure: Blood pressure cuff inflation
- Intervention group (Experimental): Remote ischemic preconditioning on the right arm is induced with a blood pressure cuff inflation at 200 mm Hg for 5 min and followed by a 5 min reperfusion at 0 mm Hg. The ischemia-reperfusion cycle is performed 3 times for a total of 30 min. This procedure is done after anesthetic induction, but before the patient is placed on cardiopulmonary bypass.
  Interventions: Procedure: Blood pressure cuff inflation

INTERVENTIONS:
Procedure: Blood pressure cuff inflation — Cuff pressure for ischemia sham is 20 mm Hg, ischemia is 200 mm Hg and reperfusion is 0 mm Hg

SUMMARY:
The study objective is to verify if a non-invasive remote ischemic preconditioning procedure (blood pressure cuff on the arm) is cardioprotective when applied before an aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned isolated aortic valve replacement (stenosis based)
* Age ≥ 18 years

Exclusion Criteria:

* Pregnancy
* Left ventricular dysfunction (LVEF< 50%)
* Myocardial Infarct (< 7days)
* Coronary artery disease (documented with >50% stenosis)
* Coronary artery bypass grafting
* Chronic renal insufficiency (creatinine >175 mmol/L or dialysis)
* Endocarditis
* Sternotomy redo
* Deep vein thrombosis to the compressed limb
* Emergency procedure
* TAVI procedure
* Planned off pump coronary artery bypass
* MAZE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-04-11 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in biochemical markers of myocardial ischemia | 6, 12, 24 and 48 hours post-operatively
  Troponin T-HS and CK-MB concentration

SECONDARY OUTCOMES:
Post-operative complications | post-operatively until 30 days
  Monitoring the safety of the strategy by monitoring post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Voisine, MD, Principal Investigator — University Laval
Locations (1):
- Hôpital Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No